CLINICAL TRIAL: NCT03423004
Title: Comparative Study of Molecular Markers in Cutaneous Inflammation Between Psoriatic Lesional Skin and Healthy Non-lesional Skin
Brief Title: Study of Molecular Markers in Cutaneous Inflammation Between Psoriatic Lesional Skin and Healthy Non-lesional Skin
Acronym: EMIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHRO-2017-12
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Psoriasis
Keywords: psoriasis; IL-22; miR-21
MeSH Terms: conditions — Psoriasis | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with lesional skin (Experimental): the sample will be taken by superficial cutaneous biopsy in psoriasic patients
  Interventions: Procedure: Biopsy
- Patients with healthy skin (No Intervention): the skin will be recovered during a surgical procedure (surgical waste) for patients who will not be opposed

INTERVENTIONS:
Procedure: Biopsy — the sample will be taken by superficial cutaneous biopsy in psoriasic patients
  Arms: Patient with lesional skin

SUMMARY:
The project topic consists on re-conciliating the fine tuners of the gene expression "microRNAs" and the immunopathogenic occasions responsible for skin disorders in context of skin infection and inflammation such as psoriasis. The skin is a network of effector cells and molecular mediators that constitute a highly sophisticated "Skin Immune System (SIS) described by Jan D Bos in 1986. The cutaneous homeostasis maintenance is dependent on the cross talk between several immune sentinels present in the different compartments of the skin as well as the interplay between innate and adaptive immune responses. The whole is under the control of gene regulation. However, cutaneous homeostasis disruption occurs when the SIS safe framework erroneously sends aggravation signals due to gene regulation disbalance via inflammatory cellular and molecular mediators into the site of infection causing chronic inflammation characterized by thick red irritated skin lesions. The latter was showed to have a characteristic microRNA (regulators of gene expression) signature.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 and 75
* Clinical diagnosis of chronic active psoriasis in non-pustular plaque
* Treated locally with topical corticosteroids

Exclusion Criteria:

* Patient who did not give express consent to participate
* No affiliation to a social security scheme
* Patient treated systemically
* Thrombocytopenic patient
* Patient known to be HIV-positive
* Septic patient
* Patient with only facial lesions
* Patient with psoriasis with joint involvement
* Patient participating in another study
* Patient protected under the law (under guardianship or trusteeship)
* Pregnant or lactating woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Increase Ratio | Day 0
  Increase ratio between relative expression of different genes (miR-21 and InterLeukin-22) of psoriatic lesional skin and non-psoriatic skin

SECONDARY OUTCOMES:
Correlation between Psoriasis Area Severity Index and miR-21 expression | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Ali ARAR, Dr, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR d'Orleans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nestle FO, Di Meglio P, Qin JZ, Nickoloff BJ. Skin immune sentinels in health and disease. Nat Rev Immunol. 2009 Oct;9(10):679-91. doi: 10.1038/nri2622. Epub 2009 Sep 18. PMID 19763149
- [Background] Finlay AY. Current severe psoriasis and the rule of tens. Br J Dermatol. 2005 May;152(5):861-7. doi: 10.1111/j.1365-2133.2005.06502.x. PMID 15888138
- [Background] Sobhan MR, Farshchian M, Hoseinzadeh A, Ghasemibasir HR, Solgi G. Serum Levels of IL-10 and IL-22 Cytokines in Patients with Psoriasis. Iran J Immunol. 2016 Dec;13(4):317-323. PMID 27999243
- [Background] Carrascosa JM, Toro Montecinos M, Ballesca F, Teniente Serra A, Martinez Caceres E, Ferrandiz C. Correlation between trough serum levels of adalimumab and absolute PASI score in a series of patients with psoriasis. J Dermatolog Treat. 2018 Mar;29(2):140-144. doi: 10.1080/09546634.2017.1341619. Epub 2017 Jul 6. PMID 28604127
- [Background] Duhen T, Geiger R, Jarrossay D, Lanzavecchia A, Sallusto F. Production of interleukin 22 but not interleukin 17 by a subset of human skin-homing memory T cells. Nat Immunol. 2009 Aug;10(8):857-63. doi: 10.1038/ni.1767. Epub 2009 Jul 5. PMID 19578369